CLINICAL TRIAL: NCT03575455
Title: The Short- And Long-Term Effects Of Submaximal Aerobic Exercise On Recovery Following Sport-Related Concussion In High School Student-Athletes
Brief Title: Sub-acute Exercise Following Sport-Related Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Tallahassee Orthopedic Clinic (Other)
Responsible Party: Principal Investigator, Phillip Worts, Principle Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF02521 - TOC
Record Dates: First submitted 2018-03-28; First posted 2018-07-02 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Sport-related Concussion
Keywords: concussion; aerobic exercise; sub-acute
MeSH Terms: conditions — Brain Concussion | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized block design using age and sex to randomize into 3 injured groups (40%, 60%, CON) and matching for 3 healthy groups (40%, 60%, CON)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Concussed participants will participate in a single 20' bout of treadmill walking at either 40% or 60% of the age-predicted HRmax.
  Healthy participants will participate in a single 20' bout of treadmill walking at either 40% or 60% of the age-predicted HRmax.
  Interventions: Behavioral: Exercise
- Seated Control (No Intervention): Concussed participants will participate in a single 20' treatment session of seated rest.
  Healthy participants will participate in a single 20' treatment session of seated rest.

INTERVENTIONS:
Behavioral: Exercise — HR-controlled treadmill walking
  Other Names: Aerobic exercise
  Arms: Exercise

SUMMARY:
Determine the safety and efficacy of sub-maximal aerobic exercise during the subacute phase of recovery following sport-related concussion.

DETAILED DESCRIPTION:
The main objective of the proposed study is to determine is exercise during the first 3-7 days following a sport-related concussion can help improve the systemic neurological dysfunction following a concussion while examining the safety and efficacy of a 20-minute, low- to moderate-intensity (40-60% of HRMAX) controlled treadmill aerobic exercise as a therapeutic modality to improve cardiovascular, psychological, vestibulo-ocular, autonomic, and cognitive function.

ELIGIBILITY:
Inclusion Criteria (concussed):

* high school student-athlete
* suffered a diagnosed concussion
* evaluated between Day 3 and Day 7 since injury

Inclusion Criteria (healthy):

* high school student-athlete
* no diagnosed concussion within the last year
* matched with concussion participant for age and gender

Exclusion Criteria:

* physical limitation prohibiting treadmill walking
* reports dizziness or lightheadedness
* presents with any contraindication for exercise participation as defined by American College of Cardiology (ACC), American Heart Association (AHA), or American College of Sports Medicine (ACSM) guidelines.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Clinical Recovery | The number of days from injury to full medical clearance up to 365 days. 80% of adolescent athletes fully recover in less than 28 days.
  Clinical recovery is defined as the duration from the time of injury to the time a patient has received full clearance without restriction.

SECONDARY OUTCOMES:
Heart rate variability (HRV) | HRV will be captured for 10 minutes before, 20 minutes during, and after 25 minutes post "treatment".
  The RR Interval will be extracted from the heart rate monitoring system.
Blood Pressure (SBP & DBP) | SBP & DBP will be captured for 10 minutes before, 20 minutes during, and after 25 minutes post "treatment".
  SBP & DBP will be recorded with an automated auscultatory BP system
Ocular Dysfunction | The King-Devick (K-D) will be administered before and within 5 minutes after the acute 20 minute "treatment"
  Improvements in ocular dysfunction will be defined as a decrease in errors or reading time
Vestibular Dysfunction | The Vestibular / Ocular Motor Screening (VOMS) will be administered before and within 5 minutes after the acute 20 minute "treatment"
  Improvements in vestibular dysfunction will be defined as a decrease in symptom provocation or pretest symptom reporting
Rating of Perceived Exertion (RPE) | RPE will be captured for 10 minutes before, 20 minutes during, and after 25 minutes post "treatment".
  Borg's CR-15 will be utilized to quantifying perceived intensity of exercise
Concussion Symptoms | Symptoms will be captured for 10 minutes before, 20 minutes during, and after 25 minutes post "treatment".
  All 22 symptoms from the Post-concussion symptom scale (PCSS) as measured on a Likert scale from 0 (not present) to 6 (severe)
Exercise Bout Completion Rates | Completion will be determined and recorded at the end of the acute 20 minute treatment.
  The rate of completion will be defined as the ability for the participant to finish the "treatment" without early termination.
Incidence of Persistent Postconcussion symptoms >28 days | The duration in days will be calculated from the day injury to the day full clearance up to 1 year.
  Persistent symptoms duration will be categorized as either ≤28 days or > 28 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Tallahassee Orthopedic Clinic, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Worts PR, Mason JR, Burkhart SO, Sanchez-Gonzalez MA, Kim JS. The acute, systemic effects of aerobic exercise in recently concussed adolescent student-athletes: preliminary findings. Eur J Appl Physiol. 2022 Jun;122(6):1441-1457. doi: 10.1007/s00421-022-04932-4. Epub 2022 Mar 18. PMID 35303160